CLINICAL TRIAL: NCT02998879
Title: A 24-month Multicenter, Open-label Phase II Trial Investigating the Safety and Efficacy of Repeated Velmanase Alfa (Recombinant Human Alpha-mannosidase) Treatment in Pediatric Patients Below 6 Years of Age With Alpha-Mannosidosis
Brief Title: Trial on Safety and Efficacy of Velmanase Alfa Treatment in Pediatric Patients With Alpha-Mannosidosis
Acronym: rhLaman-08
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-LMZYMAA1-08; 2016-001988-36 (EudraCT Number)
Record Dates: First submitted 2016-11-25; First posted 2016-12-21 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velmanase Alfa (Experimental): velmanase alfa 1mg/kg body weight infusion
  Interventions: Drug: Velmanase Alfa (e.g. Lamazym)

INTERVENTIONS:
Drug: Velmanase Alfa (e.g. Lamazym) — iv infusion treatment
  Other Names: Lamazym

SUMMARY:
The main objectives of the study are to evaluate safety and efficacy of repeated treatment with recombinant human alfa-mannosidase of patients with alfa-mannosidosis aged less than 6 years

DETAILED DESCRIPTION:
The Primary endpoints of the study include:

* Safety and tolerability of velmanase alfa as per Adverse events (AEs, including IRR), vital signs, laboratory parameters (hematology, biochemistry and urinanalysis)
* Detection of anti-velmanase alfa antibodies and neutralizing/inhibitory antibodies

The Secondary endpoints include changes from baseline to 24 months for the following parameters. Efficacy outcomes:

* Serum oligosaccharides
* Functional capacity: Peabody Developmental Motor Scale - 2nd edition (PDMS-2) scores, Mullen's Scale of Early Learning (MSEL) scores, Bruininks-Oseretsky Test Of Motor Proficiency-2nd Edition (BOT-2), when applicable by age (from 4 years) or upon the judgment of the physician
* Endurance: 3-Minute Stair Climb Test (3MSCT) and 6-Minute Walk Test (6MWT) in pediatric patients from 4 years of age, or when applicable according to the judgment of the physician, 2-Minute Walk Test (2MWT) in pediatric patients below 4 years of age, or when applicable according to the judgment of the physician
* Hearing evaluation: Otoacoustic Emissions (OAE) testing, Automatic Auditory Brainstem Response (A-ABR) audiometry
* Immunological profile, when applicable upon the judgment of the physician:
* CSF biomarkers: Tau protein (Tau), Neurofilament Protein Light (NFL), Glial Fibrillary Acidic Protein (GFAp), Oligosaccharides
* Assessment of quality of life via Questionnaire to parents
* Assessment of mannose-rich oligosaccharides in brain tissue, MRI
* Pharmacokinetic parameters

ELIGIBILITY:
Inclusion Criteria:

1. Patient's custodial parent(s) must provide signed ICF prior to the involvement of the patient in any trial-related activities
2. The subject's custodial parent(s) must have the ability to comply with the protocol
3. The subject must have a confirmed diagnosis of alpha-mannosidosis as defined by alpha-mannosidase activity in leukocytes or fibroblasts < 10% of normal activity (historical data)
4. The subject must have an age at the time of screening < 6 years.

Exclusion Criteria:

1. The subject's diagnosis cannot be confirmed by alpha-mannosidase activity < 10% of normal activity
2. Presence of known chromosomal abnormality and syndromes affecting psychomotor development, other than alpha-mannosidosis
3. History of BMT
4. Presence of known clinically significant cardiovascular, hepatic, pulmonary, or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
5. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial
6. Planned major surgery that, in the opinion of the Investigator, would preclude participation in the trial
7. Participation in other interventional trials testing the IMP within the last 3 months.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-12; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of velmanase alfa as per Adverse events | From baseline throughout study completion, at least of 2 years
  Safety and tolerability assessed as per AEs including infusion-related reactions [IRRs]
Safety and tolerability of velmanase alfa as per vital signs | From baseline throughout study completion, at least of 2 years
Safety and tolerability of velmanase alfa as per clinical laboratory parameters as per hematology | From baseline throughout study completion, at least of 2 years
Safety and tolerability of velmanase alfa as per clinical laboratory parameters as per blood biochemistry | From baseline throughout study completion, at least of 2 years
Safety and tolerability of velmanase alfa as per clinical laboratory parameters as per urinalysis | From baseline throughout study completion, at least of 2 years
Detection of anti-velmanase alfa-IgG antibodies (ADA) and neutralizing/inhibitory antibodies | From baseline throughout study completion, at least of 2 years
  Serum samples for anti-velmanase alfa-IgG antibody (ADA) testing will be obtained

SECONDARY OUTCOMES:
Evaluation of levels of Serum oligosaccharides | From baseline throughout study completion, at least for 2 years
  Assessment of change from baseline in levels of Serum oligosaccharides
Functional capacity: The Peabody Developmental Motor Scale test (PDMS-2) | From baseline throughout study completion, at least for 2 years
  Serum samples for anti-velmanase alfa-IgG antibody (ADA) testing will be obtained
Functional capacity: Bruininks-Oseretsky test of Motor Proficiency (BOT-2) when applicable by age (from 4 years) or upon the judgment of the physician | From baseline throughout study completion, at least for 2 years
Functional capacity: Mullen Scales of Early Learning (MSEL) | From baseline throughout study completion, at least for 2 years
Endurance: 3-Minute Stair Climb Test (3MSCT) in pediatric patients from 4 years of age, or when applicable according to the judgment of the physician | From baseline throughout study completion, at least for 2 years
Endurance: 6-Minute Walk Test (6MWT) in pediatric patients from 4 years of age, or when applicable according to the judgment of the physician 2-Minute Walk Test (2MWT) in pediatric patients below 4 years of age | From baseline throughout study completion, at least for 2 years
Hearing evaluation: Otoacoustic Emissions (OAE) testing | From baseline throughout study completion, at least for 2 years
Hearing evaluation: Automatic Auditory Brainstem Response (A-ABR) audiometry | From baseline throughout study completion, at least for 2 years
Immunological profile when applicable upon the judgement of the physician (Serum IgG, IgA, IgM; in vitro synthesis of IgG; in vitro proliferative response and Immunophenotype) | From baseline throughout study completion, at least for 2 years
CSF biomarkers: Tau protein (Tau) § Neurofilament Protein Light (NFL) § Glial Fibrillary Acidic Protein (GFAp) § Oligosaccharides | From baseline throughout study completion, at least for 2 years
Assessment of quality of life via Questionnaire | From baseline throughout study completion, at least for 2 years
Assessment of mannose-rich oligosaccharides in brain tissue, as measured by Magnetic Resonance Spectroscopy (MRS) | From baseline throughout study completion, at least for 2 years
Magnetic Resonance Imaging (MRI) in white matter, gray matter and in centrum semi ovale, and diffusion-MRI of the brain, | From baseline throughout study completion, at least for 2 years
Pharmacokinetic parameters to determine Cmax (Peak Concentration) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine Ctrough (Trough Plasma Concentration) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine Area Under Curve (AUC24) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine AUClast (Area Under Curve After The Last Count) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine AUCinf (Area Under Curve From Time Zero To Infinity) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine tmax (Time To Peak Concentration) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine CL (Clearance) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine t1/2 (Elimination Half-Life) | At first dose (visit 1) and after 6 months (visit 26)
Pharmacokinetic parameters to determine Rac (Obs) Observed Accumulation Ratio | At first dose (visit 1) and after 6 months (visit 26)

CONTACTS AND LOCATIONS:
Locations (6):
- Vienna, Austria
- Copenhagen, Denmark
- Lyon, France
- Germany (2):
  - Hamburg
  - Mainz
- Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-001988-36/results